CLINICAL TRIAL: NCT01790932
Title: A Phase II Trial of BKM120 in Patients With Triple Negative Metastatic Breast Cancer
Brief Title: BKM120 For Triple Negative Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Responsible Party: Principal Investigator, Nancy Lin, MD, Principal Investigator, Dana-Farber Cancer Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 12-438
Record Dates: First submitted 2013-02-07; First posted 2013-02-13 (Estimated); Results first posted 2019-01-23 (Actual); Last update posted 2019-01-23 (Actual); Status verified 2019-01

CONDITIONS: Breast Cancer
Keywords: Metastatic; Triple Negative
MeSH Terms: conditions — Breast Neoplasms; Neoplasm Metastasis | interventions — NVP-BKM120

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- BKM120 (Experimental): BKM120: 100 mg capsule once daily each day of a 28 day cycle .
  Treatment with BKM120 will continue until disease progression, unacceptable toxicity or withdrawal for other reasons.
  Interventions: Drug: BKM120

INTERVENTIONS:
Drug: BKM120
  Other Names: Buparlisib

SUMMARY:
Triple negative breast cancer (TNBC) has an aggressive phenotype and poor prognosis. This tumor type characterized by lack of expression of estrogen receptor (ER), progesterone receptor (PR) and no amplification of the human epidermal growth factor 2 (HER2) accounts for 15% of breast cancers. Limited treatment options exist in the clinic as hormonal therapies and HER2-trageted agents have proven ineffective. BKM120 is a drug that works by blocking a protein called phosphatidylinositol-3-kinase (PI3K) which may contribute to cancer growth. This drug has been used in experiments in the laboratory and information from these research studies suggests that BKM120 may help to prevent cancer cells from growing. In this research study, the investigators are looking to see if BKM120 works to stop breast cancer cells from growing.

DETAILED DESCRIPTION:
Study plan Two investigator-initiated protocols (one for US, one for Spain) will be enrolling in parallel. The first 50 participants will be recruited concurrently in US and Spain.

Stage 1 Stage 1 will include up to 50 participants with advanced TN disease. Available tumor block is required in all participants per inclusion criteria. Analysis of this tumor block will be used for correlation of predictive markers and clinical response in order to define potential subpopulation that benefit from BKM120. In Stage 1, all participants will have biopsies done at baseline, cycle 1 day 28/cycle 2 day 1 and end of treatment to analyze drug effect in the PI3K and mitogen-activated protein kinases (MAPK) pathway. This will aid to understand the pharmacodynamic effects of BKM120 in tumors with similar genetic background (triple negative disease). The enrollment of Stage 1 will ensure that at least 10 paired evaluable biopsies are obtained. After the enrollment of the first 29 evaluable subjects enrolled overall in Stage 1 (considering the US and the Spanish protocol), the Steering Committee will perform an interim analysis of safety and efficacy. If absolutely no activity is observed, the clinical trial will close and no more subjects will be enrolled. If there are early signs of activity (one patient or more achieving clinical benefit response), enrollment will proceed until 50 participants are enrolled in Stage 1. After 50 patients have been enrolled, we will analyze preliminary responses to treatment depending on the molecular status of each patient.

Stage 2 Were the trial to continue at the end of Stage 1, 50 participants would have been treated and their clinical status and response to therapy will be available. Also, paraffin blocks from these participants will have been analyzed for predictive markers of treatment effect. If there is clinical activity observed in Stage 1 and this analysis shows preliminary signs of response in a subpopulation based on the presence or absence of tumor PI3K pathway alterations, participant pre-selection may be implemented for Stage 2 (justified in an amendment before proceeding to Stage 2.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically and radiologically confirmed metastatic triple negative breast cancer
* Up to two prior lines of chemotherapy for metastatic breast cancer
* Availability of a representative tumor specimen
* At least one measurable lesion

Exclusion Criteria:

* Have received previous treatment with PI3K inhibitors
* Symptomatic central nervous system (CNS) metastases (controlled and asymptomatic CNS metastases are acceptable)
* Concurrent malignancy or has a malignancy within 3 years of study enrollment
* Any of the following mood disorders: active major depressive episode, bipolar disorder, obsessive-compulsive disorder, schizophrenia, history of suicidal attempt or ideation, homicidal ideation, greater than or equal to Common Toxicity Criteria for Adverse Events (CTCAE) grade 3 anxiety
* Concurrently using other approved or investigational antineoplastic agent and/or chemotherapy within 21 days prior to enrollment in this study
* Has received radiation therapy within 28 days prior to enrollment in this study or has not recovered from side effects of such therapy
* Major surgery within 28 days of starting therapy or has not recovered from major side effects of a previous surgery
* Poorly controlled diabetes mellitus
* History of cardiac dysfunction
* Currently receiving treatment with QT prolonging medication and the treatment cannot be discontinued or switched to a different medication
* Impairment of gastrointestinal (GI) function or GI disease that may significantly alter the absorption of BKM120
* Receiving chronic treatment with steroids or another immunosuppressive agent
* Other concurrent severe and/or uncontrolled medical condition that would contraindicate participation in this study
* History of non-compliance to a medical regimen
* Currently being treated with drugs known to be moderate or strong inhibitors or inducers of isoenzyme Cytochrome P450, family 3, subfamily A (CYP3A)
* Known history of human immunodeficiency virus (HIV)
* Pregnant or breastfeeding
* Unwilling to observe total abstinence or to use double barrier method for birth control throughout trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2012-06 (Actual); Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nancy Lin, MD, Principal Investigator — Dana-Farber Cancer Institute
Locations (4):
- United States (4):
  - Dana-Farber Cancer Institute at Faulkner Hospital, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Garrido-Castro AC, Saura C, Barroso-Sousa R, Guo H, Ciruelos E, Bermejo B, Gavila J, Serra V, Prat A, Pare L, Celiz P, Villagrasa P, Li Y, Savoie J, Xu Z, Arteaga CL, Krop IE, Solit DB, Mills GB, Cantley LC, Winer EP, Lin NU, Rodon J. Phase 2 study of buparlisib (BKM120), a pan-class I PI3K inhibitor, in patients with metastatic triple-negative breast cancer. Breast Cancer Res. 2020 Nov 2;22(1):120. doi: 10.1186/s13058-020-01354-y. PMID 33138866

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants enrolled between June 2012 and September 2014.
Period: Overall Study
Arm/Group | BKM120
Started | 50
Completed (Given treatment duration is not fixed, all participants are considered as 'Non Completed'.) | 0
Not Completed | 50
Not completed — Disease Progression | 41
Not completed — Adverse Event | 7
Not completed — Physician Decision | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Population: The analysis dataset is comprised of all enrolled participants.
Arm/Group | BKM120
Number analyzed (Participants) | 50
Age, Continuous [Median (Full Range); unit: years] | 53 [29 to 79]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 50
  Male | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 50

OUTCOME MEASURES:

1. Primary Outcome: Clinical Benefit Rate
Description: Clinical benefit rate (CBR) was defined as the proportion of participants achieving complete response (CR), partial response (PR), or stable disease (SD) for 4 months or longer based on RECIST 1.1 criteria on treatment. Per RECIST 1.1 for target lesions: CR is complete disappearance of all target lesions and PR is at least a 30% decrease in the sum of longest diameter (LD) of target lesions, taking as reference baseline sum LD. PD is at least a 20% increase in sum LD of target lesions (smallest sum LD reference), new lesions, and/or unequivocal progression of existing non-target lesions. Stable disease (SD) is defined as any condition not meeting the above criteria.
Time Frame: Disease was evaluated radiologically at baseline and every 2 cycles on treatment then every 3 months up to 2 years. Participants in this study cohort were followed for response on average approximately 2 months.
Population: The analysis dataset is comprised of all enrolled participants.
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | BKM120
Number analyzed (Participants) | 50
proportion of participants | 0.12 [0.056 to 0.238]

2. Secondary Outcome: Progression Free Survival
Description: Progression-free survival (PFS) based on the Kaplan-Meier (KM) method is defined as the duration of time from study entry to documented disease progression (PD) or death. Participants alive without PD are censored at the date of last disease assessment. Per RECIST 1.1 criteria: PD is at least a 20% increase in the sum of longest diameter (LD) of target lesions taking as reference the smallest sum LD recorded since the treatment started or the appearance of one or more new lesions. PD for the evaluation of non-target lesions is the appearance of one or more new lesions and/or unequivocal progression of non-target lesions.
Time Frame: Disease was evaluated radiologically at baseline and every 2 cycles on treatment then every 3 months up to 2 years. Participants in this study cohort were followed for PFS on average approximately 2 months.
Population: The analysis dataset is comprised of all enrolled participants.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | BKM120
Number analyzed (Participants) | 50
months | 1.8 [1.6 to 2.3]

3. Secondary Outcome: Overall Survival
Description: Overall survival (OS) is defined as the duration of time from study entry to death or date last known alive and estimated using the KM method.
Time Frame: Participants were assessed every 3 months post-treatment up to 2 years. Average survival follow-up for the study cohort was 13.8 months.
Population: The analysis dataset is comprised of all enrolled participants.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | BKM120
Number analyzed (Participants) | 50
months | 11.2 [6.2 to 25.0]

ADVERSE EVENTS:
Time Frame: Adverse events (AEs) were assessed every 2 weeks for the first 2 cycles and every cycle thereafter. Participants in this study cohort were followed for AEs on average approximately 2 months.
Description: Maximum grade toxicity by type was first calculated. Serious AEs were defined as events with treatment-attribution of possibly, probably or definitely and grade 3 or higher per Common Toxicity Criteria for Adverse Events (CTCAE) version 3. All remaining events regardless of treatment attribution were classified as Other AEs. No further data is available to specify classification of other beyond the general term.
Arm/Group | BKM120
All-Cause Mortality (participants affected / at risk) | 29/50
Serious Adverse Events (participants affected / at risk) | 17/50
Other Adverse Events (participants affected / at risk) | 44/50
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | BKM120 (N=50)
Fatigue (General disorders) | 4
Papulopustular rash (Infections and infestations) | 1
Alanine aminotransferase increased (Investigations) | 5
Aspartate aminotransferase increased (Investigations) | 4
Alkalosis (Metabolism and nutrition disorders) | 1
Anorexia (Metabolism and nutrition disorders) | 1
Hyperglycemia (Metabolism and nutrition disorders) | 2
Nervous system disorders - Other (Nervous system disorders) | 1
Dry skin (Skin and subcutaneous tissue disorders) | 1
Rash acneiform (Skin and subcutaneous tissue disorders) | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 2
Skin and subcutaneous tissue disorders - Other (Skin and subcutaneous tissue disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | BKM120 (N=50)
Anemia (Blood and lymphatic system disorders) | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 2
Blood and lymphatic system disorders - Other (Blood and lymphatic system disorders) | 1
Watering eyes (Eye disorders) | 1
Eye disorders - Other (Eye disorders) | 1
Bloating (Gastrointestinal disorders) | 1
Constipation (Gastrointestinal disorders) | 5
Diarrhea (Gastrointestinal disorders) | 9
Dyspepsia (Gastrointestinal disorders) | 2
Mucositis oral (Gastrointestinal disorders) | 5
Nausea (Gastrointestinal disorders) | 16
Rectal hemorrhage (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 2
Gastrointestinal disorders - Other (Gastrointestinal disorders) | 5
Fatigue (General disorders) | 24
Fever (General disorders) | 1
Non-cardiac chest pain (General disorders) | 2
Pain (General disorders) | 1
General disorders and administration site conditions - Other (General disorders) | 3
Hepatic failure (Hepatobiliary disorders) | 1
Allergic reaction (Immune system disorders) | 1
Papulopustular rash (Infections and infestations) | 1
Upper respiratory infection (Infections and infestations) | 1
Urinary tract infection (Infections and infestations) | 1
Infections and infestations - Other (Infections and infestations) | 2
Fracture (Injury, poisoning and procedural complications) | 1
Alanine aminotransferase increased (Investigations) | 8
Alkaline phosphatase increased (Investigations) | 1
Aspartate aminotransferase increased (Investigations) | 6
Weight loss (Investigations) | 1
Investigations - Other, specify (Investigations) | 1
Anorexia (Metabolism and nutrition disorders) | 14
Hyperglycemia (Metabolism and nutrition disorders) | 16
Hypomagnesemia (Metabolism and nutrition disorders) | 1
Hyponatremia (Metabolism and nutrition disorders) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal and connective tissue disorder - Other (Musculoskeletal and connective tissue disorders) | 2
Dizziness (Nervous system disorders) | 2
Dysgeusia (Nervous system disorders) | 2
Headache (Nervous system disorders) | 3
Peripheral sensory neuropathy (Nervous system disorders) | 3
Somnolence (Nervous system disorders) | 2
Anxiety (Psychiatric disorders) | 8
Depression (Psychiatric disorders) | 7
Insomnia (Psychiatric disorders) | 5
Libido increased (Psychiatric disorders) | 1
Psychiatric disorders - Other (Psychiatric disorders) | 7
Cystitis noninfective (Renal and urinary disorders) | 1
Hematuria (Renal and urinary disorders) | 1
Breast pain (Reproductive system and breast disorders) | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 2
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 4
Voice alteration (Respiratory, thoracic and mediastinal disorders) | 1
Alopecia (Skin and subcutaneous tissue disorders) | 1
Dry skin (Skin and subcutaneous tissue disorders) | 1
Photosensitivity (Skin and subcutaneous tissue disorders) | 1
Pruritus (Skin and subcutaneous tissue disorders) | 3
Rash acneiform (Skin and subcutaneous tissue disorders) | 5
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 3
Skin and subcutaneous tissue disorders - Other (Skin and subcutaneous tissue disorders) | 2
Hypertension (Vascular disorders) | 1
Lymphedema (Vascular disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No